CLINICAL TRIAL: NCT05498883
Title: Quality of Life Evaluation with the SRI Questionnaire of ALS Patient with Non-invasive Ventilation
Acronym: Quality EvALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP220697
Record Dates: First submitted 2022-08-11; First posted 2022-08-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; quality of life evaluation; SRI questionnaire; Zarit Burden interview
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patient requiring NIV (Other): Clinical examination, completion of the ALS-FRS score, completion of the SRI score.
  Interventions: Other: Score completion

INTERVENTIONS:
Other: Score completion — completion of the SRI score

SUMMARY:
This study aims to measure the quality of life of ALS patients by the SRI questionnaire, in two distinct patient groups : Patient requiring initiation of NIV, and patients 24 hours dependent on NIV

This study also seeks to assess the quality of life of the caregivers with the Zarit Burden interview in those two populations

DETAILED DESCRIPTION:
The course of the study is as follows:

Patient newly ventilated with NIV :

inclusion is done on the day of starting NIV. On the day of inclusion: Clinical examination, completion of the ALS-FRS score, completion of the SRI score.

For the caregiver: Completion of the Zarit Burden Inerview Reassessment of scores (SRI, Zarit-burden, ALS-FRS), at three-month and six-month follow-up

Patient dependent of NIV :

On the day of inclusion: Clinical examination, completion of the ALS-FRS score, completion of the SRI score.

For the caregiver: Completion of the Zarit Burden Inerview Reassessment of scores (SRI, Zarit-burden, ALS-FRS), at three-month follow-up

ELIGIBILITY:
Inclusion Criteria:

Patients :

* 18 years or more
* Patient followed for ALS probable or certain with Awaji criteria
* group 1 : severe chronic respiratory failure, with a decision by the attending physician to start NIV
* group 2 : complete dependence on NIV

Caregivers :

* 18 years or more
* Informed and does not object to the study
* Primary caregiver for more than 3 months of an ALS patient on NIV (either at initiation or with 24 hours NIV dependence)
* More than 30 hours spent at home per week
* Met the inclusion criteria for group 1 (NIV initiation) or group 2 (24 hours NIV dependence)

Exclusion Criteria:

Patients :

* Patient under legal protection/ guardianship
* insufficient command of French
* Severe cognitive impairment, particularly in relation to frontotemporal degeneration
* No indication criteria for NIV.

Caregivers :

* insufficient command of French
* Caregiver of a patient with another chronic pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
SRI questionnaire in patients who have indication for starting NIV | six months
  SRI questionnaire assessment at initiation of NIV, at 3-month follow-up and at 6-month follow-up

SECONDARY OUTCOMES:
SRI of patients with total ventilatory dependence in ALS | three months
  SRI questionnaire assessment at inclusion and at 3-month follow-up
Zarit burden interview in both groups | Six months
  Zarit Burden interview questionnaire in ALS patient caregiver, in both groups (initiation of NIV and NIV-dependent patients) at inclusion, 3-month follow-up (both groups) and at 6-month follow-up (in group 1)

CONTACTS AND LOCATIONS:
Overall Officials: Capucine Pr MORELOT PANZINI, MD PhD, Principal Investigator — APHP
Locations (1):
- Pneumology departement, Pitié-Salpêtrière hospital, GHU APHP-Sorbonne Université, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided